CLINICAL TRIAL: NCT06132204
Title: A Single-dose, Open-label/Pharmacokinetic and Safety Studies of HRS-7535 in Subjects With Moderate Renal Insufficiency and Healthy Subjects
Brief Title: Pharmacokinetic and Safety Studies of HRS-7535 in Subjects With Moderate Renal Insufficiency and Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shandong Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HRS-7535-102
Record Dates: First submitted 2023-11-09; First posted 2023-11-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2023-11

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HRS-7535 Tablets-Moderately renal insufficiency subjects (Experimental)
  Interventions: Drug: HRS-7535 Tablets
- HRS-7535 Tablets-Healthy subjects (Experimental)
  Interventions: Drug: HRS-7535 Tablets

INTERVENTIONS:
Drug: HRS-7535 Tablets — HRS-7535 Tablets

SUMMARY:
The study is being conducted to evaluate and compare the pharmacokinetics of HRS-7535 tablets in subjects with moderate renal insufficiency and healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Age range from 18 to 65 years old (including both ends, subject to signing the informed consent form), both male and female;
2. The subject's body weight is ≥ 50 kg, and the body mass index (BMI) is within the range of 19.0~32.0 kg/m2 (including both ends);
3. From the signing of the informed consent form until 6 months after the last administration, the subject (including partner) has no family planning and is willing to use the high-efficiency contraceptive measures specified in the plan;
4. Before the experiment, voluntarily sign an informed consent form and have a thorough understanding of the experiment content, process, and potential adverse reactions.
5. For Moderately renal insufficiency subjects， 30 mL/min ≤ GFR<60, and the renal function status is stable. Did not use drugs for treating renal insufficiency or was determined by the researcher to be stable in taking drugs for treating renal insufficiency for more than 4 weeks.
6. For Healthy subjects，90 mL/min < GFR；there was no history of chronic kidney disease during screening. Weight, age, and gender should meet the matching requirements for subjects with moderate renal insufficiency.

Exclusion Criteria:

1. During screening period, glutamate alanine aminotransferase (AST) ≥ 2 × Upper limit of normal range (ULN); Glutamate aspartate aminotransferase (ALT) ≥ 2 × ULN; Total bilirubin (TBIL) ≥ 1.5 × ULN;
2. Abnormal and clinically significant 12 lead electrocardiogram (ECG), or ECG QTcF>450 ms (corrected according to Fridericia's formula);
3. Hepatitis B surface antigen is positive, hepatitis C antibody is positive, Treponema pallidum antibody is positive, HIV antibody is positive;
4. Have a history of life-threatening diseases within 5 years (excluding basal cell skin cancer or squamous cell skin cancer);
5. Previous history of medullary thyroid cancer, multiple endocrine neoplasia type 2 or family history, previous history of pancreatitis or symptomatic gallbladder disease;
6. Previous clinical history of gastric emptying abnormalities (such as gastric outlet obstruction), severe chronic gastrointestinal diseases (such as inflammatory bowel disease and active ulcers);
7. Other clinically significant diseases (including but not limited to gastrointestinal, renal, hepatic, neurological, hematological, endocrine, tumor, lung, immune, psychiatric, or cardiovascular diseases) found within the first 6 months of screening;
8. Have undergone gastrointestinal surgery that can cause malabsorption before screening, or have taken drugs that have a direct impact on gastrointestinal peristalsis for a long time;
9. Have used drugs that may affect glucose metabolism within the first month of screening (such as systemic steroids and non-selective drugs) β Receptor blockers, monoamine oxidase inhibitors);
10. Have used glucagon like peptide peptide-1 receptor agonists within the first 3 months of screening;
11. Individuals with severe allergic diseases or known or suspected allergies or allergies to any component of the study drug (including multiple drug and food allergies);
12. Discontinuation of glucagon like peptide-1 receptor agonist therapy due to safety/tolerance reasons or lack of efficacy in the past;
13. Have received clinical trial treatment of any drug or medical device within the first 3 months or 5 half-lives (whichever is longer) before screening, or plan to participate in clinical trials of other drugs or medical devices during the trial period;
14. Screening for individuals who have consumed more than 14 units of alcohol per week within the first 6 months or who have taken alcoholic products 48 hours before administration; Or positive for alcohol breath test;
15. Smoking more than 5 cigarettes per day within the first 3 months of screening or using any tobacco products 48 hours before administration;
16. Exercise vigorously within 48 hours before administration;
17. Those who have a history of drug abuse within the past five years or have used drugs in the three months prior to the trial; Or positive for urine drug screening;
18. Donate ≥ 200 mL of blood within one month before screening; Or select trauma or surgical major surgeries who have donated blood ≥ 400 mL or lost blood ≥ 400 mL within the first 3 months;
19. Inability to tolerate venous puncture blood collection or needle dizziness;
20. Have special dietary requirements and cannot follow a unified diet;
21. Patients with fasting blood glucose>11.1 mmol/L;
22. Subjects who the researchers believe have other factors that are not suitable for participating in this experiment.
23. For Moderately renal insufficiency subjects: Have a history of kidney transplantation;Urinary incontinence or oliguria (such as<400 mL/d);Within 14 days prior to administration, medication other than those used to treat renal insufficiency and other accompanying diseases has been taken that affects the experiment; After examination and inquiry, according to the judgment of the researcher, there are serious accompanying diseases that pose a serious threat to the patient's safety or affect the patient's ability to complete this study.
24. For Healthy subjects: Have taken any medication that affects the experiment within 14 days before administration; Those who have clinical significance in judging abnormalities through comprehensive physical examination, vital signs, laboratory examination, X-ray chest X-ray, abdominal ultrasound examination, etc.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2023-12-21 (Actual); Primary Completion 2024-03-13 (Actual); Study Completion 2024-03-13 (Actual)

PRIMARY OUTCOMES:
PK parameters of HRS-7535: Cmax | 0 hour to 48 hour after administration
PK parameters of HRS-7535: AUC0-t | 0 hour to 48 hour after administration
PK parameters of HRS-7535: AUC0-inf | 0 hour to Infinity hour after administration

SECONDARY OUTCOMES:
PK parameters of HRS-7535: Tmax | 0 hour to 48 hour after administration
PK parameters of HRS-7535: t1/2 | 0 hour to 48 hour after administration
PK parameters of HRS-7535: CL/F | 0 hour to 48 hour after administration
PK parameters of HRS-7535: Vz/F | 0 hour to 48 hour after administration
Adverse events | from ICF signing date to day 7 （+3）after administration

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: Undecided